CLINICAL TRIAL: NCT00795171
Title: Randomized, Controlled Biomarker Study Evaluating the Anti-angiogenic Activity of Sunitinib in Hormone Refractory Prostate Cancer Patients Treated by Docetaxel
Brief Title: Biomarker Study for Sunitinib and Docetaxel in Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dept of Internal Medicine I, Medical University Vienna, Austria, Medical University Vienna, Austria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MK URO 4; EUDRACT 2007-003705-27
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — Docetaxel; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel + Sunitinib (Experimental): docetaxel 75mg/m2 day1 q 21d x 4 cycles, sunitinib 37.5mg/d day2 -day15 x 4 cycles
  Interventions: Drug: Docetaxel * Sunitinib
- Taxotere (Active Comparator): docetaxel 75mg/m2 day1 q 21d x 4 cycles
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel * Sunitinib — docetaxel 75mg/m2 day1 q 21d x 4 cycles, sunitinib 37.5mg/d day2 -day15 x 4 cycles
  Other Names: Taxotere + Sutent
  Arms: Docetaxel + Sunitinib
Drug: Docetaxel — docetaxel 75mg/m2 day1 q 21d x 4 cycles
  Other Names: Taxotere
  Arms: Taxotere
Drug: Docetaxel — Docetaxel 75mg/m2 q21d for 4 cycles
  Other Names: Taxotere
  Arms: Taxotere

SUMMARY:
Docetaxel and sunitinib will be compared to docetaxel for their effect on CEC/CEP spikes induced by docetaxel in HRPC patients

DETAILED DESCRIPTION:
Docetaxel (75mg/m2 q21d) is standard of care for patients with hormone refractory prostate cancer (HRPC). Recent data indicate, that chemotherapeutics given at MTD induce, besides their cytotoxic effects, mobilization of circulating endothelial cells (CEC) and - progenitors (CEP) in drug-free breaks of each cycle. In preclinical models, mobilized CEC/CEP result in tumor vasculogenesis and progression of disease.

We hypothesize that treatment with sunitinib, an anti-angiogenic tyrosine kinase inhibitor, in between 3 weekly docetaxel disrupts CEC/CEP spikes following docetaxel leading to chemosensitization and reduced tumor re-growth in HRPC patients responding to docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status of 0-2.
* Histologically proven prostate adenocarcinoma.
* All patients must have prostate adenocarcinoma that is unresponsive or refractory to androgen ablation with biochemical progression
* Measurable and/or evaluable progressive disease, which is defined by one of the following three criteria:

  * 25% increase in bidimensionally measurable soft tissue metastases
  * Appearance of new metastatic lesions (proven by CT scan, X-ray or bone scan)
  * PSA level of at least 10ng/mL, with increases on at least 2 successive occasions at least 2 weeks apart
* If the patient has been treated with antiandrogens, treatment must have been stopped at least 6 weeks prior to study randomization

Exclusion Criteria:

- prior chemotherapy for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-04 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Primary: CEC/CEP spikes induced by MTD docetaxel in patients treated with docetaxel/sunitinib relative to docetaxel monotherapy | 12 weeks

SECONDARY OUTCOMES:
Response rate and length of treatment holidays relative to docetaxel monotherapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael MK Krainer, MD, Principal Investigator — Dept of Internal Medicine I, Medical University Vienna, Austria
Locations (1):
- Dept of Internal Medicine, Vienna, Austria